CLINICAL TRIAL: NCT07386119
Title: Investigation of the Effects of Vestibular Rehabilitation and Dynamic Neuromuscular Stabilization Exercises on Balance and Mobility in Patients With Hemiplegia
Brief Title: Investigation of the Effects of Vestibular Rehabilitation and Dynamic Neuromuscular
Acronym: Dynamic
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yilmaz menek, Assoc. Prof, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-3748
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Hemiplegia; Vestibular Exercises; Physiotherapy and Rehabilitation
Keywords: Hemiplegia; Vestibular Rehabilitation; Dynamic Neuromuscular Stabilization; Balance; Mobility
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor will be masked in the assesment part in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Conventional Exercise Group (Experimental): Conventional Exercise will be conducted in this group
  Interventions: Other: Conventional Exercise programs
- Group 2: Dynamic Neuromuscular Stabilization Group (Experimental): Dynamic Neuromuscular Stabilization exercises will be done in this group
  Interventions: Other: Dynamic Neuromuscular Stabilization
- Group 3: Vestibular Rehabilitation Group (Experimental): Vestibular Rehabilitation will be conducted in this group
  Interventions: Other: Vestibular Rehabilitation Group

INTERVENTIONS:
Other: Conventional Exercise programs — This group participated in Conventional Exercise programs twice a week for six weeks.
  Arms: Group 1: Conventional Exercise Group
Other: Dynamic Neuromuscular Stabilization — This group participated in Dynamic Neuromuscular Stabilization Exercise programs twice a week for six weeks.
  Arms: Group 2: Dynamic Neuromuscular Stabilization Group
Other: Vestibular Rehabilitation Group — This group participated in Vestibular Rehabilitation programs twice a week for six weeks.
  Arms: Group 3: Vestibular Rehabilitation Group

SUMMARY:
This study will aim to investigate the effects of vestibular rehabilitation, dynamic neuromuscular stabilization (DNS), and conservative rehabilitation exercises on balance and mobility in hemiplegic patients, and to compare the exercise programs with one another. Evaluation tools include the Brunnstrom Motor Staging, Fugl-Meyer Upper Extremity Motor Function Scale, Modified Ashworth Scale, Mini-Mental State Examination, Berg Balance Scale, Stroke Impact Scale, and Timed Up and Go test.

DETAILED DESCRIPTION:
This study will aim to investigate the effects of vestibular rehabilitation, dynamic neuromuscular stabilization (DNS), and conservative rehabilitation exercises on balance and mobility in hemiplegic patients, and to compare the exercise programs with one another. A total of 45 hemiplegic patients will enrolled and randomized into three groups: Conventional Exercise Group (CEG, n = 15), Dynamic Neuromuscular Stabilization Group (DNSG, n = 15), and Vestibular Rehabilitation Group (VRG, n = 15). Each group will be participated in specialized exercise programs twice a week for six weeks. All groups will be underwent assessments before and after treatment. Evaluation tools include the Brunnstrom Motor Staging, Fugl-Meyer Upper Extremity Motor Function Scale, Modified Ashworth Scale, Mini-Mental State Examination, Berg Balance Scale, Stroke Impact Scale, and Timed Up and Go test.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Having experienced at least one stroke and presenting with hemiplegic symptoms
* Having passed at least one year since the stroke even
* Scoring at least 24 points on the Mini-Mental State Examination (MMSE)
* Being able to walk independently for at least 30 meters without assistance
* Being able to comply with and participate in the exercise program

Exclusion Criteria:

* Individuals with chronic pulmonary and/or cardiac diseases
* Presence of uncontrolled hypertension
* Conditions accompanied by peripheral nerve injury or lower motor neuron disorders
* Presence of additional neurological disorders such as ataxia, dyskinesia, or dystonia
* Severe spasticity, peripheral lesions, pressure ulcers, marked muscle atrophy, obesity, skin irritation, or use of a cardiac pacemaker
* Presence of vestibular symptoms such as vertigo or dizziness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-17 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The Fugl-Meyer Assessment of Upper Extremity | From the beginning of treatment to the end of the 6th week
  It is a standardized, stroke-specific, performance-based outcome measure used in clinical trials to evaluate motor recovery of the upper limb. It assesses movement, coordination, and reflex activity of the shoulder, elbow, forearm, wrist, and hand, providing a quantitative measure of motor impairment and recovery over time. The maximum score for the arm section is 36. During the finger-to-nose test, coordination and speed of movement are evaluated out of 6 points, while tremor, dysmetria, and speed of movement in the upper extremity are also examined in detail.
Modified Ashworth Scale (MAS) | From the beginning of treatment to the end of the 6th week
  It is a widely used clinical outcome measure in clinical trials to assess spasticity by grading the resistance encountered during passive muscle stretching. The joint is passively moved with repetitive and rapid movements, and the joint's resistance to these movements is scored.
Mini-Mental State Examination (MMSE) | From the beginning of treatment to the end of the 6th week
  It is a brief, standardized cognitive screening tool used in clinical trials to assess global cognitive function, including orientation, attention, memory, language, and visuospatial abilities. The total score ranges from 0 to 30, with higher scores indicating better cognitive performance. Scores of 24-30 indicate normal cognition, 18-23 mild cognitive impairment, and ≤17 moderate to severe cognitive impairment.
Berg Balance Scale (BBS) | From the beginning of treatment to the end of the 6th week
  This is a 14-item scale that assesses a patient's ability to maintain balance for a specific period during static and various functional movements. The scoring system ranges from 0 to 4, with 0 meaning "cannot" and 4 meaning "can do independently," and the maximum total score is 56. A total score between 0-20 indicates a high risk of falls; between 21-40 indicates a moderate risk of falls; and between 41-56 indicates a low risk of falls.
Stroke Impact Scale (SIS) | From the beginning of treatment to the end of the 6th week
  It is a stroke-specific, patient-reported outcome measure widely used in clinical trials to evaluate the perceived impact of stroke on multiple domains of health-related quality of life. Based on the obtained score, 0 indicates no recovery, whereas 100 represents complete recovery.
Timed Up and Go (TUG) | From the beginning of treatment to the end of the 6th week
  The test is a simple and widely used functional mobility assessment in clinical trials. It measures the time required for an individual to stand up from a chair, walk 3 meters, turn around, walk back, and sit down. Shorter completion times indicate better functional mobility and balance, and the test is commonly used to assess fall risk and mobility limitations.

CONTACTS AND LOCATIONS:
Overall Officials: MERVE YILMAZ MENEK, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be made available to other researchers upon reasonable request, if deemed necessary.

REFERENCES:
- [Result] Yoon HS, Cha YJ, You JSH. Effects of dynamic core-postural chain stabilization on diaphragm movement, abdominal muscle thickness, and postural control in patients with subacute stroke: A randomized control trial. NeuroRehabilitation. 2020;46(3):381-389. doi: 10.3233/NRE-192983. PMID 32250328
- See also: Effects of dynamic core-postural chain stabilization on diaphragm movement, abdominal muscle thickness, and postural control in patients with subacute stroke: A randomized control trial. NeuroRehabilitation — http://pubmed.ncbi.nlm.nih.gov/32250328/